CLINICAL TRIAL: NCT06969573
Title: The Impact of Inhaled Treprostinil on Dyspnea and Exercise Intolerance in Mild COPD; a Pilot and Feasibility Trial
Brief Title: Inhaled Treprostinil for Dyspnea and Exercise Intolerance in Mild COPD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00137313
Record Dates: First submitted 2025-04-16; First posted 2025-05-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: dyspnea; exercise tolerance; exercise capacity; inhaled Treprostinil; Prostacyclin; pulmonary vascular
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Intervention Model Description: Randomized double-blind cross-over design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants will inhale placebo (room air) from the Tyvaso Inhalation System Ultrasonic nebulizer
  Interventions: Drug: Placebo
- Treprostinil 36 mcg (Experimental): Participants will inhale 36 mcg of Treprostinil from the Tyvaso Inhalation System Ultrasonic nebulizer
  Interventions: Combination Product: Treprostinil Inhalation Solution 36 mcg
- Treprostinil 78 mcg (Experimental): Participants will inhale 78 mcg of Treprostinil from the Tyvaso Inhalation System Ultrasonic nebulizer
  Interventions: Combination Product: Treprostinil Inhalation Solution 78 mcg

INTERVENTIONS:
Drug: Placebo — Participants will breathe placebo (room air) from the Tyvaso Inhalation System Ultrasonic nebulizer
  Arms: Placebo
Combination Product: Treprostinil Inhalation Solution 36 mcg — Participants will breathe either 36 mcg of Treprostinil from the Tyvaso Inhalation System Ultrasonic nebulizer
  Arms: Treprostinil 36 mcg
Combination Product: Treprostinil Inhalation Solution 78 mcg — Participants will breathe either 78 mcg of Treprostinil from the Tyvaso Inhalation System Ultrasonic nebulizer
  Arms: Treprostinil 78 mcg

SUMMARY:
The goal of this clinical trial is to evaluate the impact of inhaled Treprostinil on breathlessness and low exercise capacity in patients living with mild chronic obstructive pulmonary disease. Participants will be asked to:

* Perform lung function and exercise tests
* Have ultrasound of their heart
* Have CT images of their lungs
* Visit the lab on 5 different occasions (plus one visit to the CT imaging clinic)

The researchers will compare the effectiveness and feasibility of inhaled Treprostinil to improve breathlessness upon exertion and exercise capacity

DETAILED DESCRIPTION:
The study consists of 6 visits (5 to the Clinical Sciences Building at the University of Alberta):

Day 1: participants will provide informed consent, medical history and health screening (Physical activity readiness questionnaire [PAR-Q+], COPD assessment test [CAT], modified medical research council [mMRC], euro quality of life- 5 dimensions [EQ-5D]), be familiarized to the laboratory and experimental measurement protocols, conduct a pulmonary function test, and conduct an incremental CPET to determine peak oxygen consumption (V̇O2peak) on the cycle ergometer. Throughout exercise, non-invasive measurements of cardiac output (impedance cardiography), heart rate (electrocardiogram), expired gases (metabolic cart), and oxygen saturation (pulse oximetry) will be completed. A small blood sample will be collected via finger prick to measure hemoglobin (to correct DLCO - part of the pulmonary function test). Ratings of perceived breathing and leg discomfort (Borg scale), as well as dimensional descriptors of dyspnea scales will be recorded throughout the exercise test, and immediately upon exercise cessation.

Days 2-4: participants will complete resting, seated, DLCO maneuvers as well as a constant workload (75% of the peak power output determined from the CPET) cycling exercise test until volitional fatigue (i.e., exhaustion) with or without inhaled Treprostinil (placebo, 36, or 78 mcg; via Tyvaso® Inhalation Solution). DLCO and its components will be evaluated by standardized multiple breath-hold technique. A small blood sample will be collected via finger prick to measure hemoglobin for the DLCO maneuvers prior to and following exercise. Throughout exercise, non-invasive measurements of cardiac output (impedance cardiography), heart rate (electrocardiogram), expired gases (metabolic cart), and oxygen saturation (pulse oximetry) will be completed. Additionally, ratings of perceived breathing and leg discomfort (Borg scale), as well as dimensional descriptors of dyspnea scales will be recorded throughout the exercise test, and immediately upon exercise cessation. The drug condition (placebo, 36, or 78 mcg) will be randomized (block randomization) by a member of our research team who is not involved in data analysis or collection.

Day 5: participants will complete supine DLCO maneuvers (multiple breath-hold technique) as well as resting echocardiography (to measure pulmonary artery and cardiac function) with and without inhaled Treprostinil (placebo, 36, and 78 mcg). A small blood sample will be collected via finger prick to measure hemoglobin for the DLCO maneuvers.

Day 6: participants will undergo a low contrast CT scan of their chest for quantification of pulmonary vascular volumes (i.e., blood vessel volume in the lungs). No drug intervention will be completed on Day 6.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild COPD (defined as having a postbronchodilator FEV1/FVC ratio <0.70 and FEV1 ≥ 80% predicted

Exclusion Criteria:

* Pre-existing heart failure and pulmonary artery hypertension.
* Known thrombocytopenia.
* Resting blood pressure of <90mmHg systolic and <50 mmHg diastolic.
* Known sensitivity to prostanoids
* Severe hepatic insufficiency

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Exercise tolerance | Within 30-45 minutes post dose
  Time to symptom limitation/exhaustion during a constant work rate test.
Exertional dyspnea | Within 30-45 minutes post dose
  Maximal perceived breathing discomfort during exercise
Ventilatory efficiency | Within 30-45 minutes post dose
  Nadir value of the ratio between ventilation and the rate of CO2 production (Ve/VCO2 nadir)

SECONDARY OUTCOMES:
Lung diffusing capacity | Within 15-30 minutes post dose
  Lung diffusing capacity (DLCO) will be measured using six-second, advanced DLCO techniques.
Pulmonary capillary blood volume (Vc) | Within 15-30 minutes post dose
  Pulmonary capillary blood volume (Vc) will be measured using six-second, advanced DLCO techniques.
Diffusing membrane Capacity (Dm) | Within 15-30 minutes post dose
  Diffusing membrane capacity will be measured using six-second, advanced DLCO techniques.
Cardiac structure and function | Within 15-30 minutes post dose
  echocardiography-derived right ventricular systolic pressure
Pulmonary vascular volumes | Day 6
  Chest computed tomography (CT) scan

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stickland, Principal Investigator — University of Alberta
Locations (1):
- Clinical Physiology Laboratory, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No